CLINICAL TRIAL: NCT04589117
Title: Expressive Writing for COVID-19 Resilience for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00105586
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Parents During COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expressive writing (Experimental): The 4-week study intervention will invite participants through a progression of expressive writing exercises designed to support emotional expression and enhance personal resilience. Weekly instruction writing sessions will be conducted via Zoom. The sessions will not be recorded, but participants who cannot attend the sessions live (or prefer not to, for any reason) will receive each week's instructions and prompts via email.
  The progression of writing exercises flows as follows:
  * Week 1: Writing to expressive difficult emotions
  * Week 2: Writing to cultivate compassion & forgiveness
  * Week 3: Writing to nurture positive emotions
  * Week 4: Writing to invite insight, perspective, & growth
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — The 4-week study intervention will invite participants through a progression of expressive writing exercises designed to support emotional expression and enhance personal resilience. Weekly instruction writing sessions will be conducted via Zoom. The sessions will not be recorded, but participants who cannot attend the sessions live (or prefer not to, for any reason) will receive each week's instructions and prompts via email.
  The progression of writing exercises flows as follows:
  * Week 1: Writing to expressive difficult emotions
  * Week 2: Writing to cultivate compassion & forgiveness
  * Week 3: Writing to nurture positive emotions
  * Week 4: Writing to invite insight, perspective, & growth

SUMMARY:
The purpose of this study is to determine the impact of a 4-week, virtually-delivered expressive writing intervention on resilience in a cohort of parents and caregivers currently navigating the COVID-19 pandemic during spring & summer of 2020.

DETAILED DESCRIPTION:
In 2016, the research team piloted a 6-week intervention on expressive writing for resilience in a population of trauma survivors. Participants self-identified as having had a recent trauma or significant life upheaval, such as a divorce, major illness, job loss, or the death of a loved one. At 6 weeks, the investigators found that participants experienced significantly improved levels of resilience and lower levels of stress, rumination, and depression. These results added to a growing body of research indicating the potential for expressive writing to be a powerful healing modality for both psychological and physical well-being.

The current COVID-19 pandemic presents the potential for trauma or significant life upheaval for nearly all members of the community and the world at large. Parents of children who are at home face unique challenges during this time. Social distancing guidelines, shelter in place protocols, school and business closures, travel restrictions, high levels of job loss, loss of childcare, and the looming threat of illness have disrupted daily routines, family life, and significantly altered life plans for many. Parents and caregivers who have unexpectedly lost childcare, are having to adjust to home schooling arrangements, and/or are having to end to heightened emotional needs in their children may experience this time as particularly difficult.

Resilience is the capacity for individuals to adapt and recover in the face of trauma, adversity, or significant sources of stress. The current collective reality magnifies the need for accessible, low-cost, effective interventions to help people cultivate resilience and other dimensions of psychological well-being.

In this study, the investigators seek to further the work the research team began in 2016 with a 4-week, virtually-delivered expressive writing intervention designed to support parents in cultivating personal resilience and emotional wellness during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

In order to have up to 40 evaluable subjects, we plan to consent up to 45 individuals. Potential subjects will be considered eligible if they are parents or primary caregivers of children aged 0-18 who have been home with them during the COVID-19 experience. Other eligibility criteria include:

* Able to speak, read, write, and understand English
* Cognitively able to provide consent
* Ability to participate in a 4-week intervention delivered via Zoom and email

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2020-08-02 (Actual)

PRIMARY OUTCOMES:
Resilience | 3 months
  Connor-Davidson Resilience Scale (CD-RISC)

SECONDARY OUTCOMES:
Perceived stress | 3 months
  Perceived Stress Scale-10 (PSS-10)
Depression symptoms | 3 months
  Center for Epidemiologic Studies Depression Scale Revised (CESDR)
Parental stress | 3 months
  Internal, non-validated questionnaire re. experience of parental stress

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Glass, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No